CLINICAL TRIAL: NCT04343482
Title: Wireless Wearable Maternal Fetal Sensors for Non-Stress Testing
Brief Title: Maternal Non-Stress Testing
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: STU00205895
Record Dates: First submitted 2020-03-30; First posted 2020-04-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: wearable vital signs sensor — vital signs monitoring during maternal non-stress testing

SUMMARY:
Percent agreement of vital signs monitoring between the experimental sensor and standard of care monitoring

ELIGIBILITY:
Inclusion Criteria:

* Maternal age >18 years old
* Pregnant mothers >26 weeks undergoing nonstress testing or delivering
* Singleton pregnancy
* No fetal abnormality or chromosomal abnormality
* Subjects willing and able to comply with requirements of the protocol
* Nurses and clinicians who will be administering the non-stress test to the pregnant subject

Exclusion Criteria:

* Women who refuse to signed the informed consent form
* Maternal age under 18 years old
* Multiple pregnancy
* Known major fetal malformation or chromosomal abnormality
* Medical or obstetric problem that would preclude the use of abdominal electrodes
* Inability to consent to this study due to medical illness, diminished intellectual capacity, or language barrier
* Women using pacemakers

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Device comparison to standard monitoring | 3 years
  The primary outcome measure is concordance of FHR tracing assessments from Rogers sensor recordings with those obtained from the current standard of care electronic fetal monitoring systems.

SECONDARY OUTCOMES:
Qualitative analyses of sensor output | 3 years
  Qualitative analyses of FHR, MHR, BP, pulse oximetry, and UC data capture from the sensors will be performed for the purpose of optimizing signal-to-noise filtering of raw data collected during the study. Any adverse events will be recorded such as skin irritation (expected to be negligible).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois, United States